CLINICAL TRIAL: NCT00890149
Title: Ondansetron for the Treatment of Heavy Drinking Among Emerging Adults
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Difficulty recruiting target sample
Sponsor: University of Maryland, Baltimore (Other)
Collaborators: National Institute on Alcohol Abuse and Alcoholism (NIAAA) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: Quadruple | Purpose: Treatment
Other Study IDs: HP-00063000; 2R01AA010522-13 (NIH)
Record Dates: First submitted 2009-04-27; First posted 2009-04-29 (Estimated); Last update posted 2023-05-26 (Actual); Status verified 2023-05

CONDITIONS: Alcohol Abuse; Alcoholism
Keywords: alcohol abuse; binge drinking; severe drinking; alcoholism; heavy drinking
MeSH Terms: conditions — Alcoholism; Binge Drinking | interventions — Ondansetron; Sugars

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Ondansetron (Experimental): Ondansetron + BASICS Plus
  Interventions: Drug: Ondansetron; Behavioral: BASICS Plus
- Placebo (Placebo Comparator): Placebo + BASICS Plus
  Interventions: Drug: Placebo; Behavioral: BASICS Plus

INTERVENTIONS:
Drug: Ondansetron — Ondansetron (4ug/kg bid),
  Other Names: Zofran
  Arms: Ondansetron
Drug: Placebo — Placebo bid
  Other Names: Sugar pill
  Arms: Placebo
Behavioral: BASICS Plus — Brief Alcohol Screening and Intervention for College Students. Brief behavioral intervention to reduce drinking.

SUMMARY:
This study will evaluate the efficacy of ondansetron + BASICS Plus in reducing severe or binge drinking among emerging adults. BASIC Plus (Brief Alcohol Screening and Intervention for College Students) has been the most validated brief intervention among college students. The BASICS program provides personal feedback, motivation, and strategies that enhance normative drinking patterns

DETAILED DESCRIPTION:
We propose to conduct a 9 week study to test the efficacy of ondansetron in a heavy drinking (non-dependent) emerging adult population. We will enroll individuals between the ages of 18 and 25 years as this period overlaps with the general population of those attending college and who can be defined as emerging adults. We will conduct a double-blind control study in which 150 individuals will be randomized into 2 groups, therefore the N will be 300.

ELIGIBILITY:
Inclusion Criteria:

* White Males and females who have given written informed consent.
* Ages 18 through 25;also, patients must weigh ≥40 kg and ≤140 kg.
* Good physical health as determined by a complete physical examination, an EKG within normal limits, and laboratory screening tests within acceptable parameters.
* At least an average of one episode of binge or heavy drinking per week in the past month prior to enrollment. For men and women, that is ≥5 and ≥4 drinks/drinking day, respectively.They also need to report at least one day of heavy drinking within the 7 days prior to randomization.
* The pregnancy test for females at intake must be negative. Additionally, women of childbearing potential must be using an acceptable form of contraception.
* Literate in English and able to read, understand, and complete the rating scales and questionnaires accurately, follow instructions, and make use of the behavioral treatments.
* Answer an advertisement in the newspaper/radio/television, and express a wish to stop heavy drinking.
* Willingness to participate in behavioral treatments to stop heavy drinking

Exclusion Criteria:

Please contact site for additional information

Ages: 18 Years to 25 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 74 (Actual)
Dates: Start 2015-09 (Actual); Primary Completion 2016-09 (Actual); Study Completion 2017-03 (Actual)

PRIMARY OUTCOMES:
Ondansetron + BASICS Plus shall be more effective at reducing severe or binge drinking among emerging adults. The treatment effect of ondansetron on reduction in severe or binge drinking shall be greatest in LL individuals. | Throughout the study
  Self-report use, Timeline Follow-back, daily drinking questionnaires, Rutgers Alcohol Problem Index, Genotyping

SECONDARY OUTCOMES:
Ondansetron adds to the therapeutic benefit of BASICS Plus, even in those with lower readiness for change | Throughout the study
  ICR Scale to abstain from using alcohol, ICR Scale for medication adherence, medication compliance,craving assessments

CONTACTS AND LOCATIONS:
Overall Officials: Bankole Johnson, DSc,MD,PhD, Principal Investigator — University of Maryland, Baltimore
Locations (1):
- Clinical Neurobehavioral Center, Columbia, Maryland, United States

IPD SHARING:
Plan to Share IPD: Undecided
A IPD sharing plan has not been developed.